CLINICAL TRIAL: NCT00132301
Title: CSP #553 - Adjuvant Therapy in Prostate Carcinoma Treatment
Brief Title: Chemotherapy After Prostatectomy (CAP) For High Risk Prostate Carcinoma
Acronym: CAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 553
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: multi-site clinical trial; prostate; radical prostatectomy; randomized
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Endpoint Committee will adjudicate evidence for progression, metastasis, and cause of death. The committee will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Docetaxel and Prednisone (Active Comparator): Chemotherapy after radical prostatectomy
  Interventions: Drug: Docetaxel; Drug: Prednisone
- Arm 2: Standard of care (No Intervention): Standard of care

INTERVENTIONS:
Drug: Docetaxel — Chemotherapy agent
  Other Names: Taxotere; Docecad
  Arms: Arm 1: Docetaxel and Prednisone
Drug: Prednisone — steroid in combination with chemotherapy agent
  Other Names: Deltasone, Orasone, Adasone, Prednisonum
  Arms: Arm 1: Docetaxel and Prednisone

SUMMARY:
VA Cooperative Study #553 is designed to prospectively evaluate the efficacy of early adjuvant chemotherapy using docetaxel and prednisone added to the standard of care for patients who are potentially cured by radical prostatectomy but who are at high risk for relapse. The standard of care is surveillance, with the addition of androgen deprivation at the time of biochemical relapse. This study will assess the effect of adding early chemotherapy to the standard of care on progression free survival in Veterans at high risk for progression after prostatectomy.

DETAILED DESCRIPTION:
VA Cooperative Study #553 is designed to prospectively evaluate the efficacy of early adjuvant chemotherapy using docetaxel and prednisone added to the standard of care for patients who are potentially cured by radical prostatectomy but who are at high risk for relapse. The standard of care is surveillance, with the addition of androgen deprivation at the time of biochemical relapse. This study will assess the effect of adding early chemotherapy to the standard of care on progression free survival in Veterans at high risk for progression after prostatectomy.

The ability of radical prostatectomy to cure prostate cancer and to therefore prevent the morbidity and mortality associated with progression to metastatic disease depends on effectively treating both local and potential systemic disease. In the United States alone, over 80,000 men per year are treated with prostatectomy to cure their disease. Because 20% of these men will be found to have locally advanced or high-grade disease, they will be at risk for relapse and morbidity from their prostate cancer. Although androgen deprivation, radiation therapy, and chemotherapy have been considered potentially effective adjuvant modalities for localized prostate cancer, there are no randomized studies that support the utility of any of these treatments as a standard of care. Ultimately, it is androgen independent prostate cancer, which causes morbidity for these patients. Docetaxel based chemotherapy has been shown to prolong survival and induce responses in up to 80% of patients with androgen independent disease, generating enthusiasm for the use of chemotherapy early in the treatment of prostate cancer. This study is designed to test the value of adjuvant chemotherapy in improving progression free survival, which is critical in preventing morbidity and mortality from relapse in patients with clinically localized, but high risk, prostate cancer.

After patients are stratified for PSA, Gleason score, tumor stage, the presence of positive margins, and the planned use of adjuvant radiation therapy, this study will randomized 300 patients from 30 VA sites, after prostatectomy, to the standard of care or to docetaxel and prednisone administered every 3 weeks for 18 weeks. Patients would then be observed with PSA for a minimum of one and a maximum of five years. The study is designed with 90% power to detect a reduction in the 5-year progression rate from 60% to 45% (15% absolute difference, 25% relative difference).

At the end of the study period (October 31, 2012), the patients in the study will continue to be passively followed for three more years. The follow-up study involved centralized remote access of the participants' medical records to obtain information on PSA levels and study endpoints.

Prostate cancer is the leading cause of malignancy for Veterans, and the second leading cause of death. Patients with high risk, localized disease account for 70% of all cancer deaths in patients treated for cure with radical prostatectomy. Effective adjuvant therapy is critical to reducing suffering and death from prostate cancer. The VA Cooperative Studies Program is uniquely placed to address this question. The VA has a longstanding history of important studies in prostate cancer, which have significantly changed the way urologic oncologists treat patients with this disease. The incidence of prostate cancer in our older, male population is substantial, the number of Veterans treated with prostatectomy continues to rise, and the incidence of high risk prostate cancer in Veterans is greater than that typically found in the community. For all of these reasons, carrying out this study within the VA through the VA Cooperative Studies Program is the optimal way to determine whether adjuvant chemotherapy will benefit men with high risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* A histologic diagnosis of cT1-T2 primary adenocarcinoma of the prostate prior to prostatectomy, with lymph node dissection at time of radical prostatectomy
* One or more of the following poor prognostic features:

  * tumor extension to seminal vesicle (pT3b) or bladder neck (T4)
  * established extracapsular extension (pT3a) and Gleason Score >= 7
  * organ confined (pT2) with positive surgical margin and Gleason 8-10
  * preoperative PSA > 20
* SWOG performance status 0-1
* PSA nadir of <= 0.1 ng/ml up to 30 days prior to randomization. Patients must be randomized within 120 days after prostatectomy.
* Laboratory values (no more than 30 days before randomization) must be as follows:

  * Absolute granulocyte count: >= 1,500/mm3
  * Platelets: >= 100,000/mm3
  * Hemoglobin: >= 10 g/dL
  * Serum Creatinine: <= 1.5 x ULN
  * AST: <= 1.5 x ULN
  * ALT: <= 1.5 x ULN
  * Serum Calcium: <= ULN
  * Total Bilirubin: <=ULN
  * Plasma Phosphorus Level: <= 6 mg/dl
* Patients with preoperative PSA > 20 ng/mL must have a negative bone scan within 120 days of randomization
* A valid, signed, and witnessed informed consent by the patient

Exclusion Criteria:

* Small cell histology
* N1 disease or M1 disease
* Clinical T3 disease prior to prostatectomy
* Any other investigational therapy
* An active serious infection or other serious underlying medical condition that would otherwise impair their ability to receive protocol treatment
* A history of cancer related hypercalcemia
* Uncontrolled heart failure
* Prior malignancy other than curatively treated squamous cell or basal cell carcinoma of the skin. If another malignancy has been treated and there is no evidence of relapse > 5 years from the time of treatment, patients are eligible
* Androgen deprivation, chemotherapy, or radiation therapy to treat prostate carcinoma
* Current peripheral neuropathy of any etiology that is greater than Grade I

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2006-06; Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lin, Study Chair — VA Puget Sound Health Care System Seattle Division, Seattle, WA; Bruce Montgomery, MD, Study Chair — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (34):
- United States (33):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, North Little Rock, Arkansas
  - VA Medical Center, Long Beach, Long Beach, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - VA Medical Center, Miami, Miami, Florida
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - VA Medical Center, Augusta, Augusta, Georgia
  - Jesse Brown VAMC (WestSide Division), Chicago, Illinois
  - VA Medical Center, Lexington, Lexington, Kentucky
  - Overton Brooks VA Medical Center, Shreveport, Shreveport, Louisiana
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center, Detroit, Detroit, Michigan
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - G.V. (Sonny) Montgomery VA Medical Center, Jackson, Jackson, Mississippi
  - VA Medical Center, Kansas City MO, Kansas City, Missouri
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Portland, Portland, Oregon
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina
  - VA Medical Center, Memphis, Memphis, Tennessee
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - Wlliam S. Middleton Memorial Veterans Hospital, Madison, Madison, Wisconsin
- VA Medical Center, San Juan, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin DW, Shih MC, Aronson W, Basler J, Beer TM, Brophy M, Cooperberg M, Garzotto M, Kelly WK, Lee K, McGuire V, Wang Y, Lu Y, Markle V, Nseyo U, Ringer R, Savage SJ, Sinnott P, Uchio E, Yang CC, Montgomery RB. Veterans Affairs Cooperative Studies Program Study #553: Chemotherapy After Prostatectomy for High-risk Prostate Carcinoma: A Phase III Randomized Study. Eur Urol. 2020 May;77(5):563-572. doi: 10.1016/j.eururo.2019.12.020. Epub 2020 Jan 8. PMID 31924316

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Chemotherapy Agent and Prednisone: Chemotherapy after radical prostatectomy
  Docetaxel: Chemotherapy agent
  Prednisone: steroid in combination with chemotherapy agent
- Arm 2: Standard of Care: Treatment by Standard of Care
Period: Overall Study
Arm/Group | Arm 1: Chemotherapy Agent and Prednisone | Arm 2: Standard of Care
Started | 141 | 157
Completed (1 participant was excluded from all analysis by the DMC) | 121 | 144
Not Completed | 20 | 13
Not completed — Death | 7 | 6
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 5 | 3
Not completed — Other | 1 | 1
Not completed — Excluded by Data Monitoring Committee | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant in Arm 1 was excluded from analysis by the Data Monitoring Committee (DMC), making the analysis population in Arm 1 140 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Chemotherapy Agent and Prednisone | Arm 2: Standard of Care | Total
Number analyzed (Participants) | 140 | 157 | 297
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 106 | 115 | 221
  >=65 years | 34 | 42 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (6.0) | 63.0 (5.3) | 62.27 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 140 | 157 | 297
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 11 | 28
  Not Hispanic or Latino | 123 | 146 | 269
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 35 | 74
  White | 94 | 113 | 207
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 9 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 140 | 157 | 297
BMI [Count of Participants; unit: Participants]
  BMI < 25 | 29 | 28 | 57
  BMI 25 to < 30 | 60 | 71 | 131
  BMI >= 30 | 51 | 58 | 109
Pre Biopsy PSA (ng/ml) [Count of Participants; unit: Participants]
  < 10 | 91 | 110 | 201
  10 to < 20 | 31 | 30 | 61
  >= 20 | 17 | 16 | 33
  Unknown or not reported | 1 | 1 | 2
Pre Prostatectomy PSA (ng/ml) [Count of Participants; unit: Participants]
  < 10 | 85 | 106 | 191
  10 to < 20 | 38 | 32 | 70
  >=20 | 17 | 19 | 36
Biopsy Gleason Score [Count of Participants; unit: Participants] — The Gleason grading system is used to help evaluate the prognosis of men with prostate cancer using samples from a prostate biopsy. Pathological scores range from 2 through 10, with higher number indicating greater risks and higher mortality.
  Participants
    <= 7 | 97 | 104 | 201
    8 to 10 | 43 | 53 | 96
Prostatectomy Gleason Score [Count of Participants; unit: Participants] — Gleason score is the grade of the tumor at prostatectomy. Scores range from 2 through 10, with higher number indicating greater risks and higher mortality. A Gleason Score of 7=3+4 means that most of the tumor is grade 3 and less is grade 4. A Gleason score of 7=4+3 means that the most of the tumor is grade 4 and less is grade 3. A Gleason score 4+3=7 tumor is more likely to grow and spread than a 3+4=7 tumor, yet not as likely as a Gleason score 8 tumor.
  Participants
    <= 7 | 7 | 4 | 11
    7: 3+4 | 52 | 60 | 112
    7: 4+3 | 35 | 36 | 71
    8-10 | 46 | 57 | 103
Clinical Stage [Count of Participants; unit: Participants] — cT stands for the clinical stage. The number is the stage of prostate cancer. The letter indicates further spreading of the cancer, such that 1<2a<2b<2c.
  Participants
    cT1 | 67 | 87 | 154
    cT2a | 36 | 28 | 64
    cT2b | 25 | 24 | 49
    cT2c | 12 | 17 | 29
    unknown or not reported | 0 | 1 | 1
Pathology Stage [Count of Participants; unit: Participants] — The T score describes how much the prostate cancer has spread within the prostate and its surrounding structures. The number is the stage of prostate cancer. The letter indicates further spreading of the cancer. The higher the score, shows the greatest risk, which is >T3b in this analysis.
  Participants
    T2a, T2b, T2c | 11 | 15 | 26
    T3a | 81 | 87 | 168
    > T3b | 48 | 55 | 103

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-Free Survival
Description: The primary objective of this study is to determine whether adding early chemotherapy based on docetaxel plus prednisone compared to standard of care alone reduces disease progression as evidenced by detectable PSA in high risk patients with prostate cancer who have undergone radical prostatectomy.
Time Frame: Up to 100 months (centralized follow-up)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Docetaxel and Prednisone | Arm 2: Standard of Care
Number analyzed (Participants) | 140 | 157
Participants | 66 | 84
Statistical Analysis 1: Comparison: Arm 1: Docetaxel and Prednisone vs Arm 2: Standard of Care; Test type: Superiority; p = 0.40, Log Rank — Log rank test stratified by site; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.58 to 1.11]

ADVERSE EVENTS:
Description: One participant in Arm 1 was excluded from analysis by the Data Monitoring Committee (DMC), making the analysis population in Arm 1 140 participants.
Groups:
- Arm 1: Chemotherapy Agent: Chemotherapy after radical prostatectomy
  Docetaxel: Chemotherapy agent
  Prednisone: steroid in combination with chemotherapy agent
Arm/Group | Arm 1: Chemotherapy Agent | Arm 2: Standard of Care
Serious Adverse Events (participants affected / at risk) | 47/140 | 50/157
Other Adverse Events (participants affected / at risk) | 79/140 | 3/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Chemotherapy Agent (N=140) | Arm 2: Standard of Care (N=157)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
Cornary artery disease (Cardiac disorders) | 3 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 3 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Spigelian hernia (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Adverse drug reaction (General disorders) | 1 | 1
Chest pain (General disorders) | 2 | 3
Death (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 2
Urinary tract infection (Infections and infestations) | 0 | 3
Clostridial infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 3 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Accident at work (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Traumatic arthritis (Injury, poisoning and procedural complications) | 1 | 0
Biopsy bone (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Hyperglcaemia (Metabolism and nutrition disorders) | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cartoid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral vascular accident (Nervous system disorders) | 1 | 2
Hemmorhage intracranial (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 1
Mayasthenia gravis (Nervous system disorders) | 0 | 1
Thalamic infarction (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 1 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Achohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Biopolar disorder (Psychiatric disorders) | 1 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 3 | 5
Urinary retention (Renal and urinary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 3
Organic erectile dysfunction (Reproductive system and breast disorders) | 0 | 2
Chronic obtructive pulonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulomary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Vasculitic rash (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic bypass (Surgical and medical procedures) | 0 | 1
Lipoma excision (Surgical and medical procedures) | 0 | 1
Chemotherapy (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 2 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1
Arterial Thrombosis (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Chemotherapy Agent (N=140) | Arm 2: Standard of Care (N=157)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 55 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 3 | 0
White blood cell count decreased (Investigations) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 25 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Carpal tunnel decompression (Surgical and medical procedures) | 0 | 1
Hernia repair (Surgical and medical procedures) | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes